CLINICAL TRIAL: NCT06098313
Title: Efficacy and Safety of Allogeneic Hematopoietic Cell Transplantation Using Post-transplantation Cyclophosphamide for Graft-versus-host Disease Prophylaxis in Higher-risk Myelodysplastic Syndrome, Chronic Myelomonocytic Leukemia, and Secondary AML Patients
Brief Title: HCT With PTCy in Higher-risk MDS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Je-Hwan Lee, M.D. Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRMDS_PTCy_2019
Record Dates: First submitted 2023-10-19; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Patients With MDS, Acute Myeloid Leukemia (AML) Evolving From MDS, and Chronic Myelomonocytic Leukemia (CMML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PTCy (Experimental): Patients who receive post-transplantation cyclophosphamide
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide — -Cyclophosphamide 50 mg/kg/day i.v. daily on days 3 and 4 (for 2 days)

SUMMARY:
This study is conducted to evaluate the efficacy of post-transplantation cyclophosphamide with myeloablative or reduced-intensity conditioning regimen for allogeneic hematopoietic cell transplantation (HCT) in patients with higher-risk myelodysplastic syndrome (MDS). The efficacy of the treatment will be measured in terms of the GVHD-free, relapse-free survival.

The secondary end points of the study include engraftment, relapse incidence, non-relapse mortality, graft-versus-host disease, donor chimerism, immune reconstitution, infections, and survivals (overall and event-free).

DETAILED DESCRIPTION:
This study is conducted to evaluate the efficacy of post-transplantation cyclophosphamide with myeloablative or reduced-intensity conditioning regimen for allogeneic hematopoietic cell transplantation (HCT) in patients with higher-risk myelodysplastic syndrome (MDS). The efficacy of the treatment will be measured in terms of the GVHD-free, relapse-free survival.

The secondary end points of the study include engraftment, relapse incidence, non-relapse mortality, graft-versus-host disease, donor chimerism, immune reconstitution, infections, and survivals (overall and event-free).

ELIGIBILITY:
Inclusion Criteria:

* MDS defined by WHO classification, CMML, or AML evolving from MDS A. International Prognostic Scoring System (IPSS) > 1.0 or bone marrow blast ≥ 5% at any time points before HCT or B. AML progressed from MDS or C. CMML with bone marrow blast ≥ 5% at any time points before HCT
* Patients receiving first HCT
* Patients with appropriate hematopoietic cell donors A. HLA-matched sibling donor B. Unrelated donor C. HLA-mismatched familial donor
* 15 years old or older , under 75 years
* Adequate performance status (Karnofsky score of 70 or more)
* Adequate hepatic function (AST or ALT < 3 x upper normal limits and bilirubin < 1.5 x upper normal limit).
* Adequate renal function (creatinine < 2.0 mg/dL or creatinine clearance ≥ 50 mL/min)
* Adequate cardiac function (left ventricular ejection fraction ≥ 50% on heart scan or echocardiogram)
* Adequate pulmonary function: DLCO, FEV1, and FVC ≥ 45% predicted by pulmonary function tests
* Signed and dated informed consent must be obtained from both recipient and donor.

Exclusion Criteria:

* Presence of significant active infection
* Presence of uncontrolled bleeding
* Any coexisting major illness or organ failure
* Patients with psychiatric disorder or mental deficiency severe as to make compliance with the treatment unlike, and making informed consent impossible
* Nursing women, pregnant women, women of childbearing potential who do not want adequate contraception
* Patients with a diagnosis of prior malignancy unless disease-free for at least 5 years following therapy with curative intent (except curatively treated nonmelanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia)
* Presence of contraindications to cyclophosphamide (patients receiving pentostatin, symptomatic cystitis, urinary tract obstruction, with a history of hypersensitivity reactions to the component of the drug)

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 113 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
GVHD-free, relapse-free survival | 8 years
  This study is conducted to evaluate the efficacy of post-transplantation cyclophosphamide with myeloablative or reduced-intensity conditioning regimen for allogeneic hematopoietic cell transplantation (HCT) in patients with higher-risk myelodysplastic syndrome (MDS). The efficacy of the treatment will be measured in terms of the GVHD-free, relapse-free survival.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided